CLINICAL TRIAL: NCT02905669
Title: Measurement of Contractile Activity and Distensibility of the Esophago-gastric Junction, of the Esophagus and of the Pylorus: Normal Values in Controls Under General Anesthesia (NormaFLIP Study)
Brief Title: Normal Values for Esophageal and Pyloric Impedance Planimetry Under General Anesthesia (NormaFLIP)
Acronym: NormaFLIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0457
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Dysfunction; Pylorus Dysfunction
Keywords: distensibility; impedance planimetry; esophagus; esophago-gastric junction; pylorus
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoFLIP (Experimental): Esophago-gastric junction distensibility will be assessed in patients thanks to impedance planimetry using EndoFLIP device.
  Interventions: Device: EndoFLIP

INTERVENTIONS:
Device: EndoFLIP — Esophago-gastric junction distensibility will be assessed in patients thanks to impedance planimetry using EndoFLIP device

SUMMARY:
Impedance planimetry using Endoscopic Functional Lumen Imaging Probe (EndoFLIP) device is a promising diagnostic tool to assess esophageal, esophago-gastric junction and pylorus function. It allows the measurement of esophageal and pylorus distensibility as well as contractile activity in response to distension. Examination is useful performed under sedation. General anesthesia might affect distensibility values. The aim of this study is to normal values for esophageal, esophago-gastric junction and pylorus distensibility in controls during an upper gastro-intestinal endoscopy performed under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Subject older than 18 years and younger than 80 years
* Subject referred for upper gastro-intestinal endoscopy under general anesthesia for anemia, intestinal metaplasia in the stomach, Helicobacter pylori screening, or submucosal dissection
* Subject with health insurance
* Written informed consent

Exclusion Criteria:

* Patient younger than 18 years or older than 80 years
* Pregnancy or breast feeding
* Previous history of esophago-gastric surgery or vagotomy
* Previous history of Parkinson disease or diabetes mellitus
* Contra-indication to upper gastro-intestinal endoscopy
* Esophageal varices
* Esophageal diameter smaller than 5 mm
* Contra-indication to general anesthesia
* Hiatal hernia greater than 3 cm on endoscopy
* Esophageal or gastric cancer otherwise than superficial lesion with indication of submucosal dissection
* Typical symptoms (heartburn, regurgitation) of gastro-esophageal reflux disease and/or gastroesophageal reflux disease (GERD)-Q score greater or equal to 8
* Nausea, vomiting or epigastric pain
* Dysphagia with Sydney score greater ou equal to 50
* Incapability to give consent
* No written informed consent
* Participation to another study at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
Esophago-gastric junction distensibility | The day of gastro-intestinal endoscopy

SECONDARY OUTCOMES:
Esophageal distensibility | The day of gastro-intestinal endoscopy
Pylorus distensibility | The day of gastro-intestinal endoscopy
Esophageal contractile activity in response to distension | The day of gastro-intestinal endoscopy
  distension volume for presence of esophageal repetitive contraction
Side effects occurence | The day of gastro-intestinal endoscopy
  Occurrence of pain, aspiration and vomiting
Side effects occurence | The day after gastro-intestinal endoscopy
  Occurrence of pain, aspiration and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Exploration Fonctionnelle Digestive, Hôpital Edouard Herriot, Lyon, France